CLINICAL TRIAL: NCT06300983
Title: Effectiveness of a Psychoeducational Intervention on Myositis Patients' Quality of Life and Well-Being: A Randomized Controlled Trial
Brief Title: Effectiveness of a Psychoeducational Intervention on Myositis Patients' Quality of Life and Well-Being
Acronym: HRQoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR(AG)398/2022
Record Dates: First submitted 2024-02-12; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Quality of Life; Myositis
Keywords: Clinical trial; Inflammatory myopathy; Myositis; Psychoeducational intervention; Health related quality of life
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): The intervention consisted of 5 sessions, with each lasting 100 minutes and delivered on a weekly basis.
  Interventions: Behavioral: Psychoeducative
- Control group (Placebo Comparator): The control group, which do not receive any psychoeducative intervention
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Psychoeducative — The intervention consiste of 5 sessions (Table 1), with each lasting 100 minutes and delivered on a weekly basis. Individual meetings will be conducted with each participant prior to starting the group work. These were considered pre-intervention sessions, during which patients provided informed consent to participate in the study and the first assessment tests were administered.
  Arms: Experimental group
Behavioral: Placebo — The control group, which do not receive any psychoeducative intervention
  Arms: Control group

SUMMARY:
Purpose. Myositis is a rare disease associated with impaired health-related quality of life. A study evaluating the effectiveness of an intervention to improve the quality of life and well-being of myositis patients is presented.

Materials and Methods. All myositis patients in a health district are contacted. Eligible patients are randomly assigned to the experimental or control group. A psychoeducational intervention of 5 100-min sessions focusing on the disease as related to daily life is conducted only in experimental patients. Several reliable tools to measure quality of life and well-being are administered twice, before and after the intervention, to both groups.

DETAILED DESCRIPTION:
Materials and methods The Medical Research Ethics Committee and Research Projects Commission of the Vall d'Hebron University Hospital approved the project [number PR(AG)398/2022]. Attending to circumstances of the intervention and to enhance methodological quality, the study is designed as a randomized controlled trial with a control group and an experimental group, with two measurement time points. The CONSORT statement is followed to conduct the study.

Participants Patients are eligible for enrolment based on the following inclusion criteria.

1. a definite diagnosis of myositis according to the International Myositis Classification Criteria (score > 90) and
2. the ability to understand the purpose and procedures of the study, and motivation and agreement to participate.

A large cohort of adult myositis patients attending our outpatient clinic (Systemic Autoimmune Diseases Unit of Vall d'Hebron General Hospital, Barcelona, Spain) are potential candidates for the study. Vall d'Hebron General Hospital is a 700-bed referral and teaching hospital for a catchment population of nearly 450,000 inhabitants. Virtually all patients from the area with suspected myositis are referred to Vall d'Hebron, where they are diagnosed, treated, and followed up, whether the disease is severe or not.

All candidate patients are contacted by telephone and invited to participate in the study during a 2-month period. Patients are excluded from the study if they do not meet the diagnostic criteria or are hospitalized for an extremely severe illness, declined to participate, required excessive convincing for participation, deemed likely to play a disruptive role in the group, are younger than 18 years, had severe psychiatric conditions, or had an unfavourable short-term prognosis.

Psychoeducational Intervention The psychoeducational program will be carried out in the experimental group during a two-month period. Control patients do not participate in the intervention, and are treated as usual, and placed on a waiting list to receive the psychoeducational intervention after completion of the study. Patients who receive the intervention had no contact with the control participants. The intervention consists of 5 sessions, with each lasting 100 minutes and delivered on a weekly basis. Individual meetings are conducted with each participant prior to starting the group work. These are considered pre-intervention sessions, during which patients provided informed consent to participate in the study and the first assessment tests is administered.

Two specialized professionals participate in the group sessions: a leader and an external observer present during the process. The leader positioned herself within the group ecology, facilitating the dynamics and development of the sessions. The observer, located outside the group ecology, but in the same room, is responsible for preparing complete minutes of each session and detailed observations, recording the topics discussed and the session structure, as well as presences, absences, delays, and critical incidents, among other relevant data.

The duration and structure of each session is constant, with an introduction phase of 30 minutes, a central phase (the most substantial part of each session) of 50 minutes, and a final phase of 20 minutes. The methodological approach used in the study allow for systematic and consistent implementation of the group psychoeducational program. The combination of individual and group sessions, together with the presence of an external observer, provide a comprehensive view of the progression of the participants and the topics covered.

Measures

Participants are required to fill out a series of questionnaires related with the objectives of the study at 2 time points: before the start of the intervention and on the last day of the intervention. The control group, which do not participate in the intervention, filled out the same questionnaires at the same 2 time points. The battery of questionnaires included the following scales:

World Health Organization Quality of Life Measure (WHOQOL-BREF): a comprehensive, generic questionnaire designed to evaluate various aspects of quality of life. The WHOQOL-BREF consists of 26 items, with 24 items covering four domains: physical health, psychological health, social relationships, and environment. Additionally, 2 global questions inquire about overall quality of life and satisfaction with health. Participants rated each item on a 5-point scale, in which higher scores indicate better quality of life. The assessment was based on the experiences of the past 2 weeks. Results from the 4 domains multiplied by 4 gives a score from 0 to 100, with higher scores indicating better quality of life.

The Spanish version of the WHOQOL-BREF has demonstrated good psychometric properties among elderly Spanish individuals, validating its suitability for the study population.

World Health Organization Well-Being Index (WHO-5): a five-item scale used to assess positive well-being experienced over the past 2 weeks. Each item is rated on a 6-point Likert scale, ranging from 0 (indicating at no time) to 5 (representing all of the time). The total score ranges from 0 to 25. The total multiplied by 4 gives a score from 0 to 100, with higher scores indicating a greater sense of well-being. The WHO-5 has shown high reliability [18].

Self-Efficacy to Manage Chronic Disease Scale (Spanish version, SEMCD-S): developed and validated to assess self-management following an intervention conducted in Stanford University's Chronic Disease Self-Management Program. The questionnaire comprises 4 items, and participants rate each item on a scale from 1 (very unsure) to 10 (very sure). The self-efficacy value is determined as the average of the 4 scores obtained. Higher scores on the scale indicates higher levels of self-efficacy. The questionnaire has shown favorable psychometric properties, indicating good reliability.

International Physical Activity Questionnaire - Short Form (IPAQ) (validated Spanish short-form version). This questionnaire assesses types of physical activity according to their intensity levels and the amount of time spent sitting, as individuals engage in their daily routines. These factors are used to estimate the total physical activity in MET-minutes per week and the duration of sitting time. The tool includes inquiries about 3 types of activity-walking, moderate-intensity activities, and vigorous-intensity activities-performed over the last 7 days, along with a question about sitting time. The overall physical activity (PA) score is obtained by summing up the MET-minutes per week for all 3 types of activities. The study classifies the population into 3 PA levels-low, moderate, and high-following the IPAQ guidelines. Test-retest reliability has indicated good stability.

Participant information encompassed sociodemographic data, which comprised age, sex, marital status, household composition, educational background, and employment status. Clinical data, such as age at diagnosis, specific diagnosis, and years of disease follow-up, were also recorded.

Statistical analysis SPSS version 28 (SPSS Software Inc., Chicago, IL) is used for the statistical analyses. The McNemar test is carried out for nominal dependent variables, and repeated measures ANOVA are used for quantitative variables [22]. Eta squared is used as a measure of effect size. Effect size values around 0.01 are considered a small effect, around 0.06 a medium effect, and around 0.14 a large effect.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of myositis according to the International Myositis Classification Criteria (score > 90)
* Ability to understand the purpose and procedures of the study, and motivation and agreement to participate.

Exclusion Criteria:

* Do not meet the diagnostic criteria
* Patients hospitalized for an extremely severe illness
* Patients who declined to participate
* Patients who required excessive convincing for participation
* Patients who deemed likely to play a disruptive role in the group
* Patients younger than 18 years
* Patients who had severe psychiatric conditions or had an unfavorable short-term prognosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 2 months
  WHOQOL-The WHOQOL-BREF consists of 26 items, with 24 items covering four domains: physical health, psychological health, social relationships, and environment. Additionally, 2 global questions inquire about overall quality of life and satisfaction with health. Participants rated each item on a 5-point scale, in which higher scores indicate better quality of life. The assessment was based on the experiences of the past 2 weeks. Results from the 4 domains multiplied by 4 gives a score from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Albert S Selva-O'Callaghan, Prof, Principal Investigator — Vall d'Hebron General Hospital
Locations (1):
- Hospital Universitari Vall d'Hebron. Universitat Autonoma de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Armadans-Tremolosa I, Palacin-Lois M, Castrechini-Trotta A, Sanduvete-Chaves S, Chacon-Moscoso S, Selva-O'Callaghan A. Effectiveness of a psychoeducational intervention on myositis patients' quality of life and well-being: a randomized controlled trial. Orphanet J Rare Dis. 2024 Nov 1;19(1):411. doi: 10.1186/s13023-024-03426-0. PMID 39487522